CLINICAL TRIAL: NCT06625034
Title: Randomized Phase III Trial of Rapid-Plan Knowledge-Based Planning vs. Human-Driven Planning for Prostate Cancer Radiotherapy
Brief Title: Radiation Therapy With RapidPlan Knowledge-based Planning vs Human-Driven Planning for Treatment of Prostate Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMROA2451; NCI-2024-07870 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-006449 (Other: Mayo Clinic Institutional Review Board); GMROA2451 (Other: Mayo Clinic Radiation Oncology)
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; Photons; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm A (human-driven treatment planning, radiation therapy) (Active Comparator): Patients receive human-driven treatment planning and undergo radiation therapy over 15-30 minutes on 5-44 fractions per standard of care. Additionally, patients undergo MRI pre-treatment and blood sample collection and PET throughout study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Radiation: Photon Beam Radiation Therapy; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Radiation Therapy Treatment Planning and Simulation
- Arm B (RapidPlan treatment planning, radiation therapy) (Experimental): Patients receive RapidPlan treatment planning and undergo radiation therapy over 15-30 minutes on 5-44 fractions per standard of care. Additionally, patients undergo MRI pre-treatment and blood sample collection and PET throughout study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Radiation: Photon Beam Radiation Therapy; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Radiation Therapy Treatment Planning and Simulation

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Radiation: Photon Beam Radiation Therapy — Undergo radiation therapy
  Other Names: External beam radiation therapy using photons (procedure); Photon; Photon EBRT; Photon External Beam Radiotherapy; PHOTON Therapy; Radiation, Photon Beam
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy Treatment Planning and Simulation — Receive human-driven treatment planning
  Other Names: Radiation Therapy Treatment Planning/Simulation
  Arms: Arm A (human-driven treatment planning, radiation therapy)
Radiation: Radiation Therapy Treatment Planning and Simulation — Receive RapidPlan treatment planning
  Other Names: Radiation Therapy Treatment Planning/Simulation
  Arms: Arm B (RapidPlan treatment planning, radiation therapy)

SUMMARY:
This phase III trial compares the effects of radiation therapy using RapidPlan, trademark, knowledge-based planning to human-driven planning in treating patients with prostate cancer. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill tumor cells and shrink tumors. Successful delivery of radiation requires planning to develop a treatment plan for how and where the radiation is to be delivered. RapidPlan is a knowledge-based treatment planning tool that automatically creates an optimal treatment plan based on identified targets and organs at risk for radiation exposure. Human-driven treatment planning by a dosimetrist, the current standard of care, requires significant resources and time and may vary within and among radiation centers. Giving radiation therapy with RapidPlan knowledge-based planning may have similar or less side effects compared to human-driven planning in treating patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if RapidPlan knowledge-based planning is non-inferior to human-driven planning regarding treatment-related rates of grade 3 or higher genitourinary (GU) and gastrointestinal (GI) adverse events at 3 months post-radiotherapy for prostate cancer.

EXPLORATORY OBJECTIVES:

I. After completion of radiation therapy, determine the incidence of:

Ia. Grade 2 or greater GU and GI toxicity at 3 months (Common Terminology Criteria for Adverse Events [CTCAE] version 5); Ib. Quality of life 3 months post-radiotherapy; Ic. Rate of achieving dose-volume constraints. II. Determine if there are any statistical differences in dose-volumes results with RapidPlan knowledge-based planning.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A (HUMAN-DRIVEN): Patients receive human-driven treatment planning and undergo radiation therapy over 15-30 minutes on 5-44 fractions per standard of care. Additionally, patients undergo magnetic resonance imaging (MRI) pre-treatment and blood sample collection and positron emission tomography (PET) throughout study.

ARM B (KNOWLEDGE-BASED): Patients receive RapidPlan treatment planning and undergo radiation therapy over 15-30 minutes on 5-44 fractions per standard of care. Additionally, patients undergo MRI pre-treatment and blood sample collection and PET throughout study.

After completion of study treatment, patients are followed up at 3 and 12 months then yearly for up to year 5.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years old
* Histologically confirmed prostate cancer
* Clinical or pathologic stages T1c-T3b, Nx or N0-1, M0-1 (American Joint Committee on Cancer [AJCC] criteria 8th edition [Ed])
* Planned definitive dose radiotherapy to the prostate or prostate bed
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 assessed within 90 days of enrollment
* Patients must sign Institutional Review Board (IRB) approved study specific informed consent
* Patients must complete all required pre-entry tests within the specified time frames
* Patients must be able to start treatment (radiation) within 180 days of study registration
* In case of confusion about the eligibility or ineligibility of an individual patient, the principal investigator (PI) can be used as the arbiter and a note to file will be added to the subject's regulatory binder to document outcome

Exclusion Criteria:

* Previous pelvic radiation > 5 Gy
* Planned delivery of radiotherapy to pelvic lymph nodes
* Planned delivery of brachytherapy of the prostate
* Active rectal diverticulitis, Crohn's disease affecting the rectum, or ulcerative colitis (non-active diverticulitis and Crohn's disease not affecting the rectum are allowed)
* Prior hip replacement or penile implant
* Major medical, addictive, or psychiatric illness which in the investigator's opinion, will prevent the consent process, completion of the treatment and/or interfere with follow-up. (consent by legal authorized representative is not permitted for this study)
* Indwelling or intermittent urinary catheter use

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-02-02 (Actual); Primary Completion 2028-05-28 (Estimated); Study Completion 2033-05-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3 or higher genitourinary (GU) and gastrointestinal (GI) adverse events (AEs) | Up to 3 months post-radiotherapy
  AEs will be defined using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Comparisons between treatment arms will be made using a non-inferiority test for the difference between two proportions with an alpha level of 5%. The proportion of patients experiencing grade 3 or higher GU or GI AEs over the number of patients eligible for toxicity will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Y. Yu, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials